CLINICAL TRIAL: NCT03336411
Title: Personalized Technology-Supported Counseling to Reduce Glycemic Response in Dietary Weight Loss: The Personal Diet Study
Brief Title: A Personalized Diet Study to Reduce Glycemic Exposure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: American Heart Association (Other); Weizmann Institute of Science (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-00741
Record Dates: First submitted 2017-11-06; First posted 2017-11-08 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Pre-diabetes; Overweight and Obesity
MeSH Terms: conditions — Glucose Intolerance; Overweight; Obesity | interventions — Telemedicine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mHealth (Active Comparator)
  Interventions: Behavioral: Personalized mHealth
- Personalized mHealth (Experimental)
  Interventions: Behavioral: mHealth

INTERVENTIONS:
Behavioral: mHealth — Behavioral weight loss intervention using behavioral counseling focusing on physical activity and a one-size-fits-all, calorie-restricted, diet.
  Arms: Personalized mHealth
Behavioral: Personalized mHealth — Behavioral weight loss intervention with personalized dietary recommendations based on machine learning algorithm that integrates gut microbiota, dietary intake, physical activity and various blood parameters to predict postprandial glycemic response.
  Arms: mHealth

SUMMARY:
The aim of this 2-phase, randomized clinical trial will be to examine the effects of two behavioral weight loss interventions on weight loss. This study will be conducted in 200 overweight or obese prediabetic individuals recruited from community-based settings.. Phase 1 will include 6-months of active intervention. Phase 2 will consist of 6-months of maintenance and observation. Measurements will occur at screening, baseline, 3, 6, and 12 months. Participants will be randomized with equal allocation to 2 groups: (1) a standardized behavioral weight loss intervention with a one-size-fits-all regimen that includes counseling about restriction of calories and calories from fat, and physical activity, delivered using mHealth technology, or (2) all of the elements of mHealth, plus personalized dietary recommendations to minimize glycemic response to meals. Participants will be required to attend 6 separate visits over both phases of the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy overweight or obese prediabetic (HbA1c <8.0%)
* BMI ≥27 kg/m2
* Oral medications with metformin, sulfonylureas, DPP4 inhibitors
* Posses smartphone or use study loaner smartphone

Exclusion Criteria:

* unable or unwilling to provide informed consent
* unable to participate meaningfully in an intervention that involves self-monitoring using software available in English (e.g., due to uncorrected sight impairment, illiterate, non-English-speaking, dementia)
* unwilling to accept randomization assignment
* women who pregnant, or plan to become pregnant in the next 13 months, or who become pregnant during the study
* institutionalized (e.g., in a nursing home or personal care facility, or those who are incarcerated and have limited control over diet)
* unwilling to delay bariatric surgery for the next 12 months
* diagnosed with heart disease, kidney disease, or retinopathy, (to rule-out those with long-standing T2D)
* chronically active inflammatory or neoplastic disease in the past 3 years
* diagnosed with a chronic gastrointestinal disorder (e.g. inflammatory bowel disease or celiac disease)
* diagnosed with active infection requiring antibiotics in the last 3 months or who develop an active infection requiring antibiotics during the study
* taking medications containing acetaminophen and are unwilling or unable to discontinue its use during the study (acetaminophen affects the accuracy of the continuous glucose monitoring [CGM] device)
* taking chronic immunosuppressive medications or used them in the 3 months prior to participation, or during the study
* managing glycemia with insulin, GLP-I agonists (exenatide, liraglutide, lixisenatide, albiglutide, dulaglutide), insulin secretagogues (Glimepiride, Glipizide, Glyburide, Repaglinide, Nateglinide), or SGLT2 inhibitors (canagliflozin, dapagliflozin, empagliflozin, empagliflozin/metformin, dapagliflozin/metformin)
* prescribed medications expected to result in weight loss such as Orlistat, Naltrexone, Bupropion, Lorcaserin, Phentermine, Topiramate, or Liraglutide, and who are unwilling to delay treatment with these medications for the next 12 months
* +/- 5% weight change within last month at screening
* a eGFR <60 mL/min/1.73m2
* younger than 18 or older than 80 years old.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-10-27 (Actual)

PRIMARY OUTCOMES:
Body weight, percent change | 6 months
  the primary outcome will be relative weight change as a percentage of body weight at baseline and 6-months using calibrated scale.

SECONDARY OUTCOMES:
Body Composition | 6 & 12 months
  the secondary outcome will be absolute and relative changes in fat and lean body mass based on bioelectrical impedance analysis (BIA) from baseline to 6-months, 6-months to 12-months and baseline to 12-months
Metabolic Adaptation | 6 & 12 months
  the secondary outcome will be the change in resting metabolic rate overall, and in relation to body weight and lean body mass from baseline to 6-months, 6- to 12-months, and baseline to 12-months. Resting metabolic rate will be estimated using indirect calorimetry with the participant in a fasting state (12 hours)
Weight regain | 12 months

OTHER OUTCOMES:
Glycemic variability (GV ) | 6 months
  GV will be obtained from continuous glucose monitoring (CGM) tracings collected with the Abbott FreeStyle Libre Pro.
RAGE/AGE/S100/A8/A9 | 6 & 12 MONTHS
  In the first 30 participants randomized to the study (15 in each group) having BMI ≥35 kg/m2, at each measurement time point we will examine activation of the RAGE/AGE/S100A8/A9 pathway using measurements of sRAGE, AGE level by ELISA, levels of S100A8/A9 by ELISA, circulating TNF-alpha, IL1-beta, IL4, IL10, and IL-17
Adipokines | 6 & 12 months
  Leptin and high molecular weight adiponectin each measurement time point in the subsample of participants having BMI ≥35 kg/m2
Self-efficacy | 3,6, 12-months
  Self-efficacy for weight loss will be assessed using the well-validated Weight Efficacy Lifestyle Questionnaire (WEL)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Ann Sevick, ScD, Principal Investigator — NYU Langone Medical Center, Department of Population Health; Eran Segal, PhD, Principal Investigator — Weizmann Institute of Science, Department of Computer Science and Applied Mathematics
Locations (1):
- New York University School of Medicine, New York, New York, United States

REFERENCES:
- [Derived] Berube LT, Wang C, Curran M, Pompeii ML, Hu L, Barua S, Li H, St-Jules DE, Schoenthaler A, Segal E, Bergman M, Popp CJ. Personalized dietary feedback mediates the association of dietary self-monitoring adherence and weight loss: a post-hoc analysis of the Personal Diet Study. J Nutr. 2026 Jan 13:101364. doi: 10.1016/j.tjnut.2026.101364. Online ahead of print. PMID 41539436
- [Derived] Kharmats AY, Popp C, Hu L, Berube L, Curran M, Wang C, Pompeii ML, Li H, Bergman M, St-Jules DE, Segal E, Schoenthaler A, Williams N, Schmidt AM, Barua S, Sevick MA. A randomized clinical trial comparing low-fat with precision nutrition-based diets for weight loss: impact on glycemic variability and HbA1c. Am J Clin Nutr. 2023 Aug;118(2):443-451. doi: 10.1016/j.ajcnut.2023.05.026. Epub 2023 May 24. PMID 37236549
- [Derived] Popp CJ, Hu L, Kharmats AY, Curran M, Berube L, Wang C, Pompeii ML, Illiano P, St-Jules DE, Mottern M, Li H, Williams N, Schoenthaler A, Segal E, Godneva A, Thomas D, Bergman M, Schmidt AM, Sevick MA. Effect of a Personalized Diet to Reduce Postprandial Glycemic Response vs a Low-fat Diet on Weight Loss in Adults With Abnormal Glucose Metabolism and Obesity: A Randomized Clinical Trial. JAMA Netw Open. 2022 Sep 1;5(9):e2233760. doi: 10.1001/jamanetworkopen.2022.33760. PMID 36169954
- [Derived] Popp CJ, Zhou B, Manigrasso MB, Li H, Curran M, Hu L, St-Jules DE, Aleman JO, Vanegas SM, Jay M, Bergman M, Segal E, Sevick MA, Schmidt AM. Soluble Receptor for Advanced Glycation End Products (sRAGE) Isoforms Predict Changes in Resting Energy Expenditure in Adults with Obesity during Weight Loss. Curr Dev Nutr. 2022 Mar 29;6(5):nzac046. doi: 10.1093/cdn/nzac046. eCollection 2022 May. PMID 35542387
- [Derived] Popp CJ, Butler M, Curran M, Illiano P, Sevick MA, St-Jules DE. Evaluating steady-state resting energy expenditure using indirect calorimetry in adults with overweight and obesity. Clin Nutr. 2020 Jul;39(7):2220-2226. doi: 10.1016/j.clnu.2019.10.002. Epub 2019 Oct 14. PMID 31669004
- [Derived] Popp CJ, St-Jules DE, Hu L, Ganguzza L, Illiano P, Curran M, Li H, Schoenthaler A, Bergman M, Schmidt AM, Segal E, Godneva A, Sevick MA. The rationale and design of the personal diet study, a randomized clinical trial evaluating a personalized approach to weight loss in individuals with pre-diabetes and early-stage type 2 diabetes. Contemp Clin Trials. 2019 Apr;79:80-88. doi: 10.1016/j.cct.2019.03.001. Epub 2019 Mar 4. PMID 30844471